CLINICAL TRIAL: NCT02603874
Title: The Development of a Vertebra Localizing Aid Medical Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Target Tape (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H15-02787
Record Dates: First submitted 2015-11-05; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Spinal Cord Neoplasms; Spinal Fractures
Keywords: Fluoroscopy; Spinal Fusion; Wrong Level Surgery
MeSH Terms: conditions — Spinal Cord Neoplasms; Spinal Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Target Tape (Experimental): Including target tape in the procedure
  Interventions: Device: Target Tape
- Control (No Intervention): Without target tape in the procedure

INTERVENTIONS:
Device: Target Tape — Comparing procedures using Target Tape against procedures not using Target Tape
  Arms: Target Tape

SUMMARY:
The current method of incision localization in many surgical procedures requires a doctor to reference a medical image, such as an X-ray, to judge where on the body an incision should be made. However, the precise information of the scan is not shown on the patient's skin. Surgeons commonly use palpation to locate the point of incision. They may feel for the area directly or find landmarks under the skin and estimate the location from there. This can be challenging due to the difficulty of feeling and distinguishing each vertebra, especially for new surgeons, since palpation is a skill derived through experience.

If palpation proves ineffective, they may be forced to use fluoroscopy. By referencing the fluoroscopy image the surgeon moves a radiopaque marker, such as their surgical tool, closer to the area of interest. Fluoroscopy is time-consuming, and exposes medical personnel and the patient to radiation. Many fluoroscopic images may be required in a single procedure. The purpose of this study is to test the efficacy and benefits of a new medical device that will aid in radiological localization. The hypothesized outcome would be smaller incisions, faster localization and a reduction in fluoroscopy use.

By identifying the efficacy of this new medical device, "Target Tape", there is the potential outcome of making smaller incisions, faster localization, a reduction in fluoroscopy use and a reduced chance in surgical error and the associated costs.

Target Tape is a non invasive device that is in a grid format that is placed against the subject's skin. The grid pattern will then appear on the medical imaging scan. The medical practitioner can correlate device grid on the body to the medical scan image to make their incisions in more accurate locations.

DETAILED DESCRIPTION:
Consent must first be obtained from the prospective patient before Target Tape can be incorporated into the procedure. When a target procedure is scheduled to occur, the surgeon will first determine if Target Tape would be appropriate to use. The procedure will need to be able to integrate Target Tape into it using the Method of Use described above. The decision to then pursue the procedure will be under the discretion of the medical practitioner and consent from the patient. Depending on the procedure, the medical practitioner may need to communicate to the OR or the radiology department to integrate Target Tape into their protocol, since the practitioner making the incisions(s) may not always be the one applying it. Examples of spine procedures that may utilize Target Tape may be stabilization of fractures, tumor removals, fusions, discectomies and kyphoplasties. . Once the procedure is determined to be appropriate to accommodate Target Tape, the medical practitioner will approach the prospective patient and explain how the device will be utilized, the benefits and potential risks associated with it, and answer any questions the patient may have. A representative from Target Tape Inc may be on hand to aid with this process and may also observe said procedure to record the necessary information. The consent form will then be signed and Target Tape will then be utilized during the procedure.

The methodology of creating an outcome measure will occur over 2 stages with multiple steps in each stage:

Stage I: Proof of Concept

1. Specify measurement goals
2. Proof of Concept Testing
3. Item generation
4. Item reduction

Stage 2: Verification 5. Verification Testing 6. Reliability 7. Validity 8. Interpretability

(i) Subjects (ii) Involved Groups (iii) Data Collection (iv) Statistics

Stage 1: Proof of Concept

1. Measurement goals

   The specific measurement goals are to verify specific procedures that benefit from Target Tape. This serves as primary evidence, beyond the initial feedback and opinions of medical professionals. Based on the benefits to the procedures, significant performance variables will be determined that can be measured in Stage 2 testing. The significant performance variables may be either qualitative or quantitative:
   * Ease of use (surgeon opinion)
   * Usefulness (surgeon opinion)
   * Time analysis
   * Incision length
   * Fluoroscopy use

   Other variables that may need to be collected are certain subject characteristics (ie. age, gender, height, weight and skin pigmentation). These variables help control for the effects of variable skin characteristics that may affect the performance of Target Tape.

   Based upon interviews with medical professions such as surgeon and radiologists, initial target procedures include stabilization of fractures, tumor removals, fusions, discectomies and kyphoplasties.

   This research is intended to be a multi participant study and may include a variety of different spine physicians who are interested in utilizing the device in their procedures. The overall method of use and testing remains consistent between the various participants.
2. Proof of Concept Testing When a target procedure is scheduled to occur, the surgeon will first determine if Target Tape would be appropriate to use. The procedure will need to be able to integrate Target Tape into it using the Method of Use described above. The decision to then pursue the procedure will be under the discretion of the medical practitioner and consent from the patient. Depending on the procedure, the medical practitioner may need to communicate to the OR or the radiology department to integrate Target Tape into their protocol, since the practitioner making the incisions(s) may not always be the one applying it. Once the procedure is determined to be appropriate to accommodate Target Tape, the medical practitioner will approach the prospective patient and explain how the device will be utilized, the benefits and potential risks associated with it, and answer any questions the patient may have. The consent form will then be signed and Target Tape will then be utilized during the procedure.
3. Variable generation Item generation will be conducted in two stages. First, a list of items will be created from the current outcome. The items will be grouped according to the domains of: ease of use, device limitations, patient characteristics, time analysis, incision length and fluoroscopy use. Second, this list will be distributed to the surgeons/medical practitioners who have used the device and any missing items will be included. It is anticipated that up to 10 procedures would have used the device.
4. Variable reduction The list of items generated in the step above will be administered to doctors who will be asked to rate the items according to importance. Any items that are deemed insignificant will be removed from the list. The objective of the item reduction step is to find variables that are important to patients, doctors, and the hospital. Furthermore, a definitive list of target procedures will be chosen, with procedures of no observed benefits taken off the list.

   Stage 2: Verification
5. Verification Testing Subject to the testing results of Stage 1, there will be a set of significant performance variables determined for each respective target procedure. The significant variables may include time in the OR, incision length and fluoroscopy exposure. The purpose of Stage 2 would be to verify the significant variables for each procedure. Exclusion criteria would be created based upon the outcome of Stage 1. Target Tape would then be randomly utilized in the procedures, with controls for who is performing the procedure and patient characteristics (such as gender, age, weight, height and skin pigmentation). Observation of the significant performance variable occurs for all the procedures. The significant variables may be highly dependent upon the medical practitioner; therefore, the sample size will be related to the number of procedures the respective practitioner performs in a given amount of time. Stage 2 may not be a necessary step for the initial development of Target Tape; due to the simplicity of the device as well as qualitative factors, the cost-benefit analysis may not necessarily require a lengthy statistical study.
6. Reliability Reliability refers to the consistency of the tool; the tool being the criteria and testing to measure the significant performance variables. The device that will be used will be the same design throughout Stage 2.
7. Validity Validity refers to how well an instrument (i.e. criteria and testing) measures what it claims to measure. The different types of validity are: face, content, construct and criterion validity. Face validity ensures that the significant performance variables make sense and will be ensured throughout the creation of the criteria by involving surgeons, radiologists and patients. Content validity is the extent to which an instrument covers a representative sample of the domain in question. Again this will be ensured during the creation of the tool by involving surgeons, radiologists and patients. Construct validity assesses the factors that can affect ratings. Construct validity will also be assessed by looking for floor and ceiling effects. Criterion validity may be assessed, and is the extent to which the utilization of Target Tape is predictive of surgical outcomes (i.e. incision lengths, radiation exposure, and procedure times).
8. Interpretation Quantitative measurements are measured on an absolute scale: incision lengths measured in millimeters, procedure times in seconds, and fluoroscopy exposure in the number of 'shots' as well as the time of live exposure in seconds (if possible). Controls for patient characteristics will be recorded in absolute values, i.e. 37 years, 5'8" 160 lbs. In the interpretation and analysis, these controls may be grouped. There are also measures of the surgeon's opinion on the qualitative 'ease of use' and qualitative 'usefulness'. This would be a of 10, with the 10 mark representing the best possible score. In this case, zero would be difficult to use or can see no usefulness, respectively. These scores would be converted into percentages. They can be interpreted to find relative usefulness across various surgical procedures, as well as the effects of independent variables (i.e. physical controls).

   (i) Subjects The population for which Target Tape is designed for is an individual undergoing a medical procedure in which a medical imaging scan is utilized to assist with incision localization. These medical imaging scans may include X-ray, fluoroscopy, CT or MRI. Depending on the nature of the procedure, the scan(s) may be done preoperative or intraoperative. The surgeon may use the scan image in conjunction with palpation to determine the incision site. Examples of possible procedures include stabilization of fractures, tumor removals, fusions, discectomies and kyphoplasties. Although the above conditions represent procedures that can occur in patients of any age, the population to which this study will be directed is those who would not be allergic to any medical adhesives, medical skin inks, and/or copper metal.

   The designated surgeon or medical practitioner will carry out subject recruitment at an appropriate time before preoperative imaging or before the operation. Those who agree may be asked to complete the consent form at that same time.

   Sample size

   Stage 1:

   1-2 Spinal surgeons up to 10 patients

   The number of medical practitioners in each type of procedure may fluctuate. The number of patients may vary depending on the relative magnitude of the observations and feedback from the medical practitioners.

   Stage 2:

   The sample sizes for each segment of this stage corresponds to sample sizes used to create outcome measures in the different populations. After Stage 1 has been completed, the sample sizes for Stage 2 will be assessed and a statistical model will be created at that time. A preliminary estimate would require 5 times the sample size of per procedure of Stage 1 to be a sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Surgical spine procedures involving the use of medical imaging to determine the vertebra site (ex. fusions, tumor removals, fracture repairs, discectomies). The medical imaging scans may include planar X-rays, fluoroscopy, CT or MRI scans
* Able and willing to consent

Exclusion Criteria:

* Subjects who may have allergies to medical skin adhesives

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in Fluoroscopy Exposure | 6 months
  Measuring the decreased amount of fluoroscopy radiation exposed to the medical staff and the patient

CONTACTS AND LOCATIONS:
Overall Officials: Jin W Tee, MD, FRACS, Principal Investigator — University of British Columbia

REFERENCES:
- [Background] Kim KD, Li W, Galloway CL. Use of a radiopaque localizer grid to reduce radiation exposure. Ann Surg Innov Res. 2011 Aug 9;5:6. doi: 10.1186/1750-1164-5-6. PMID 21827694